CLINICAL TRIAL: NCT00138723
Title: A Phase 3, Parallel Group, Randomized, Double-Blind, Placebo Controlled Multicenter Trial to Investigate the Efficacy, Tolerability and Safety of Fesoterodine Sustained Release in Subjects With Overactive Bladder Syndrome
Brief Title: Trial to Investigate the Efficacy, Tolerability and Safety of Fesoterodine Sustained Release in Subjects With Overactive Bladder Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SP584
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

INTERVENTIONS:
Drug: SPM 907

SUMMARY:
This Phase 3 trial will investigate the efficacy, tolerability and safety of fesoterodine fumarate (SR) (fesoterodine; SPM 907) in adult male and female subjects with overactive bladder syndrome. The trial is a randomized, double-blind placebo controlled multicenter trial.

The trial consisted of a 2 week Run-In period, 12 week double-blind Treatment period and 2 week Safety Follow-Up period. Subjects were randomized to one of 3 treatment arms receiving either fesoterodine fumarate 4mg, fesoterodine fumarate 8mg, or placebo during the double-blind Treatment period.

Two primary efficacy variables will be assessed for submission in the United States: change in the average number of micturitions (frequency) per 24 hours and the change in the average number of urge incontinence episodes per 24 hours. For the submissions in the European Union, the first primary variable will be the change in the average number of micturitions (frequency) per 24 hours and the co-primary variable is the treatment response, based on a treatment benefit scale. All continuous variables will be measured as changes from baseline to value after 12 weeks of treatment. The following safety variables were observed and assessed: adverse events, change in residual urinary volume (mL), change in laboratory parameters, change in vital signs, change in electrocardiogram (ECG), change in physical examination and change in urological/urogynecological examination.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder syndrome

Exclusion Criteria:

* Less than 8 micturitions in 24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- [Derived] Cardozo L, Khullar V, El-Tahtawy A, Guan Z, Malhotra B, Staskin D. Modeling dose-response relationships of the effects of fesoterodine in patients with overactive bladder. BMC Urol. 2010 Aug 19;10:14. doi: 10.1186/1471-2490-10-14. PMID 20723260
- [Derived] Staskin D, Michel MC, Nitti V, Morrow JD, Wang J, Guan Z. Efficacy of fesoterodine over 24 hours in subjects with overactive bladder. Curr Med Res Opin. 2010 Apr;26(4):813-8. doi: 10.1185/03007990903585707. PMID 20121659